CLINICAL TRIAL: NCT04167839
Title: Effects of Sensory Diets on a Child's Sensory Processing Skills, Psychosocial Skills, and Classroom Engagement
Brief Title: Effects of Sensory Diets on Children's Sensory Processing Skills, Psychosocial Skills, and Classroom Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pingale, Vidya, OTR (Individual)
Collaborators: Tina S. Fletcher, EdD, MFA, OTR (Unknown); Catherine Candler, PhD, OTR (Unknown); Noralyn Pickens, PhD, OT (Unknown); Karen Dunlap, EdD (Unknown)
Responsible Party: Principal Investigator, Pingale, Vidya, OTR, Doctoral Student, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TWU protocol# 19711
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Sensory Processing Disorder; Special Education; Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Second observers were masked from participants' evaluation data and treatment phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sensory diet — Sensory diets are one of the interventions occupational therapists use in school-based settings to manage manifestations of sensory processing disorder. Sensory diets are composed of exercises and multisensory activities that are tailored for children and provide them sensorimotor experiences to facilitate their participation in daily activities.
  Other Names: Non-therapeutic activities or activities without a therapeutic goal (Placebo)

SUMMARY:
This study investigated the effects of a sensory diet intervention program on five children with a sensory processing disorder. The effect was investigated on children's sensory processing skills, psychosocial skills, and classroom engagement.

DETAILED DESCRIPTION:
Sensory diets are one of the interventions occupational therapists use in school-based settings to manage manifestations of sensory processing disorder. However, very few studies have investigated the effectiveness of sensory diets, and the results of these studies were mixed. Past studies also had methodological limitations. Therefore, this study investigated the effect of sensory diets on children's sensory processing skills, psychosocial skills, and engagement in classroom activities. This study used a single-subject ABCA design. Five children between the ages of five and eleven years participated in the study. The study consisted of an initial baseline phase A1, the control intervention phase B, sensory diets intervention phase C, and the second baseline phase A2. Each phase lasted for seven days. The PI videotaped each participant for fifteen minutes each school day during all phases to collect the data. The participants were videotaped during classroom group activities. Visual analysis of the data showed that sensory diets had a positive effect on participants' sensory processing, psychosocial skills, and classroom engagement.

ELIGIBILITY:
Inclusion Criteria:

- Children between the ages of four and eleven years and attending pre-kindergarten through fourth grade

* Children eligible for occupational therapy services under the special education eligibility criteria or under section 504 of the Rehabilitation Act of 1973-subpart D. This subpart of section 504 ensures children with disabilities who do not meet the eligibility criteria for special education services and are placed in general education classrooms receive the necessary support and related services (such as occupational therapy) to fully participate in general education classrooms.
* Children who scored in the Definite Difference range (+ 2 SD) or Probable Difference (+ 1 SD) ranges on two or more sections or quadrants on the Sensory Profile-2, Teacher Questionnaire (SP-2 Teacher Questionnaire; Dunn, 2015) were included in this study

Exclusion Criteria:

Children with medical concerns, such as cardiac conditions, posing risk to participate in resistive (strenuous) gross motor activities or children who used mobility devices were excluded from the study as these conditions may have hindered their participation in sensory diet activities.

* Children who were on medications, such as stimulants, anti-anxiety or anti-convulsive medications were excluded from the study as these medications may influence the clinical representation of SPD and interfere with the study outcomes.
* Children who were currently receiving sensory diets or received sensory diets six months prior to the beginning of the study were excluded from the study to control for confounding.

Ages: 4 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Change in frequency of a target behaviors related to psycho-social behaviors | The data was collected for 28 days; each day for each phase for 15 minutes.
  This outcome measure was individualized for each participant and detected change in frequency of psycho-social behaviors. The target behavior was identified and individualized based on the analysis of the intake data using classroom observations, Sensory profile school companion 2nd edition results, Behavior assessment system for children 3rd edition results, and teacher interview.
Change in duration of a target behavior related to off-task behaviors. | The data was collected for 28 days; each day for each phase for 15 minutes.
  This outcome measure individualized for each participant and detected change in duration of off-task behaviors. The target behavior was identified and individualized based on the analysis of the intake data using classroom observations, Sensory profile school companion 2nd edition results, Behavior assessment system for children 3rd edition results, and teacher interview.
Change in duration of a target behavior related to sensory seeking behaviors. | The data was collected for 28 days; each day for each phase for 15 minutes.
  This outcome measure individualized for each participant and detected change in duration of sensory seeking behaviors. The target behavior was identified and individualized based on the analysis of the intake data using classroom observations, Sensory profile school companion 2nd edition results, Behavior assessment system for children 3rd edition results, and teacher interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Vidya Pingale, Cliffside Park, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fazlioglu Y, Baran G. A sensory integration therapy program on sensory problems for children with autism. Percept Mot Skills. 2008 Apr;106(2):415-22. doi: 10.2466/pms.106.2.415-422. PMID 18556898
- [Background] Lopez, M., & Swinth, Y. (2008). A group proprioceptive program's effect on physical aggression in children. Journal of Occupational Therapy, Schools & Early Intervention, 1(2), 147-166. doi: 10.1080/19411240802313044
- [Background] Case-Smith J, Weaver LL, Fristad MA. A systematic review of sensory processing interventions for children with autism spectrum disorders. Autism. 2015 Feb;19(2):133-48. doi: 10.1177/1362361313517762. Epub 2014 Jan 29. PMID 24477447
- [Background] Watling R, Hauer S. Effectiveness of Ayres Sensory Integration(R) and Sensory-Based Interventions for People With Autism Spectrum Disorder: A Systematic Review. Am J Occup Ther. 2015 Sep-Oct;69(5):6905180030p1-12. doi: 10.5014/ajot.2015.018051. PMID 26356655
- [Result] Devlin S, Healy O, Leader G, Hughes BM. Comparison of behavioral intervention and sensory-integration therapy in the treatment of challenging behavior. J Autism Dev Disord. 2011 Oct;41(10):1303-20. doi: 10.1007/s10803-010-1149-x. PMID 21161577